CLINICAL TRIAL: NCT05526326
Title: OrganOx Metra® New Enrollment Post-Approval Study
Brief Title: OrganOx Metra® New Enrollment PAS
Status: Completed | Type: Observational
Sponsor: OrganOx Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: P200035/PAS003
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; Normothermic perfusion; Biliary complications
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Post-Approval Transplant Recipient cohort: Adult liver transplant recipients who are transplanted with an OrganOx metra® perfused DBD or DCD donor liver according to the approved indication and matching eligibility criteria
  Interventions: Device: Transplant with normothermic machine perfused (NMP) donor liver

INTERVENTIONS:
Device: Transplant with normothermic machine perfused (NMP) donor liver — The enrolled recipient will receive a DBD or DCD donor liver that underwent normothermic machine perfusion with the OrganOx metra®
  Other Names: OrganOx metra® normothermic machine perfusion

SUMMARY:
The objective of the OrganOx metra® New Enrollment Post-Approval Study is to collect data on the post-transplant clinical outcomes of DBD and DCD donor livers preserved and assessed on the OrganOx according to the current indications for use in the real-world setting.

DETAILED DESCRIPTION:
The OrganOx metra® New Enrollment Post-Approval Study is a multi-site, single arm, unblinded post-approval study that will enroll deceased DBD or DCD donor liver and adult liver transplant recipients according to the current indication and that match the eligibility criteria below.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or greater
* Subject is registered as an active recipient on the UNOS waiting list for liver transplantation
* Subject, or legally authorized representative, is able and willing to give informed consent and HIPAA authorization
* Subject is able and willing to comply with all study requirements (in the opinion of the Investigator)

Exclusion Criteria:

* Subject requiring all of the following at the time of transplantation:

  1. Oxygen therapy via a ventilator/respirator
  2. Inotropic support
  3. Renal replacement therapy
* Subject has acute/fulminant liver failure (UNOS status 1A)
* Subject planned to undergo simultaneous transplantation of more than one organ (e.g., liver and kidney) from the same liver donor
* Subject is pregnant (as confirmed by urine or serum pregnancy test) or nursing
* Concurrent enrollment in another clinical study. Subjects enrolled in clinical studies or registries where only measurements and/or samples are taken (no test device or test drug) are allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult primary liver transplant candidates on the waiting list for liver transplant at a U.S. liver transplant center and who meet the eligibility criteria at the participating study centers
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Adverse biliary-related events | 12-months post-transplant
  Adverse biliary-related events as measured by biliary complications

SECONDARY OUTCOMES:
Graft survival | 12-months post-transplant
  Liver graft survival post-liver transplant as measured by the number of subjects needing a re-transplant
Subject survival | 12-months post-transplant
  Subject survival post-liver transplant

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Loyola University, Maywood, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Mount Sinai, New York, New York
  - Duke University, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided